CLINICAL TRIAL: NCT01572025
Title: Efficacy of Dehydroepiandrosterone to Overcome the Effect of Ovarian Aging - A Pilot Double Blinded Randomised Controlled Trial
Brief Title: Dehydroepiandrosterone (DHEA) Intervention To Treat Ovarian Aging
Acronym: DITTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11054; 2011-002425-21 (EudraCT Number)
Record Dates: First submitted 2012-03-19; First posted 2012-04-05 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Infertility; Ovarian Aging; Diminished Ovarian Reserve (DOR); Predicted Poor-responders
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHEA supplementation (Experimental)
  Interventions: Drug: Dehydroepiandrosterone
- Control (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dehydroepiandrosterone — Dehydroepiandrosterone (DHEA)(St Mary's Pharmaceutical Unit Cardiff and Vale) DHEA 75 mg capsule. 1 capsule taken once daily for at least 12 weeks prior commencing ovarian stimulation protocol
  : Stimulation protocol standard long down-regulation protocol, using human menopausal gonadotropin (HMG)
  Arms: DHEA supplementation
Drug: Placebo — Matched Placebo containing no active ingredient. 1 capsule taken once daily for at least 12 weeks prior commencing ovarian stimulation protocol
  : Stimulation protocol standard long down-regulation protocol, using human menopausal gonadotropin (HMG)
  Arms: Control

SUMMARY:
* To test the hypothesis that supplementation of DHEA for at least twelve weeks prior to and during ovarian stimulation increases oocyte quantity (number of oocytes retrieved) and oocyte quality (clinical pregnancy rates and molecular markers) following IVF and IVF/ICSI treatment.
* To evaluate the feasibility of conducting a large multicentre trial

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the role of DHEA in counteracting the effects of ovarian ageing in an in-vitro fertilization (IVF) model. The study will examine whether the use of DHEA could improve clinical pregnancy rates following IVF treatment in women predicted to have aged ovaries by increasing oocyte quantity (ovarian response to gonadotrophins) and/ or by improving oocyte quality. The oocyte quality will be assessed by morphological and molecular markers.

This study will provide a mechanistic framework for translational research on mechanisms of ovarian ageing and drug interventions to slow down the ovarian ageing process and subsequent adverse physical and psychological consequences. Further, the data that will be produced from this research will have the potential to influence clinical practice in fertility clinics worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Women aged above 23 years with diminished ovarian reserve (predicted to be poor-responder), defined as antral follicle count <10 and/or Anti-Mullerian hormone <5pmol/L
* Women undergoing IVF and IVF/ICSI treatment
* Women must have a regular spontaneous menstrual cycle of 21 - 35 days

Exclusion Criteria:

* Women with BMI >35 Kg/M2
* Women with a single ovary
* Women with untreated hydrosalpinx/ submucous fibroid/ endometrial polyp at the start of treatment
* Women with any history of seizure disorders
* Women with previous participation in this trial in an earlier treatment cycle
* Women with any known endocrine disorders such as congenital adrenal hyperplasia, thyroid diseases, hyperprolactinemia
* Known allergy to DHEA
* Diabetic women on insulin as insulin lowers DHEA levels and might reduce the effectiveness of DHEA supplements.

Ages: 23 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | within 15 weeks after DHEA/Placebo supplementation
  Oocytes retrieved within 15 weeks after DHEA/placebo supplementations.
Feasibility to conduct a large multicentre randomised controlled trial | with in 20 weeks of the research period (per participant)
  Feasibility is evaluated by assessing recruitment rates and compliance of the recruited participants with DHEA/ placebo intake and follow up rates

SECONDARY OUTCOMES:
Oocyte quality (clinical and molecular markers) | The sample is collected at 14-16 weeks after recruitment and assessment is performed at one year.
  Clinical pregnancy rates (Pregnancy rate determined at week 5 to 7 after embryo transfer).
  Molecular markers of oocyte quality as assessed by expression of cumulus cell molecular markers of oocyte competence and also by assessing energy consumption (pyruvate, lactate and glucose utilization) from the media by the oocytes and embryos (nutritional finger printing)
Aneuploidy rates in the immature oocytes and unfertilized oocytes using microarray technology | The sample is collected at 14-16 weeks after recruitment and assessment is performed at one year.

CONTACTS AND LOCATIONS:
Overall Officials: Kannamannadiar Jayaprakasan, MRCOG,PhD., Principal Investigator — Division of Obstetrics and Gynaecology, School of Clinical Sciences, University of Nottingham; Bruce Campbell, PhD, DSc, Study Director — University of Nottingham; Nick Raine-Fenning, MRCOG, PhD, Study Director — University of Nottingham
Locations (1):
- Nottingham University Research and Treatment Unit in Reproduction (NURTURE), Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Derived] Jayaprakasan K, Narkwichean A, Maalouf WE, Campbell BK. Efficacy of dehydroepiandrosterone to overcome the effect of ovarian ageing (DITTO): a proof of principle randomised controlled trial protocol. BMJ Open. 2014 Oct 8;4(10):e005767. doi: 10.1136/bmjopen-2014-005767. PMID 25296654